CLINICAL TRIAL: NCT04467047
Title: Safety and Feasibility of Allogenic Mesenchymal Stromal Cells in the Treatment of COVID-19
Brief Title: Safety and Feasibility of Allogenic MSC in the Treatment of COVID-19
Acronym: COVID19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200148
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Sars-CoV2
Keywords: Mesenchymal Stromal Cells; COVID-19; Sars-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intravenous 1*10E6 MSCs/kg body weight Mesenchymal Stromal Cells infusion
  Interventions: Biological: Mesenchymal Stromal Cells infusion

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells infusion — Intravenous 1*10E6 MSCs/kg body weight Mesenchymal Stromal Cells infusion

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is spreading worldwide and has become a public health emergency of major international concern. Currently, no specific drugs or vaccines are available. For severe cases, it was found that aberrant pathogenic T cells and inflammatory monocytes are rapidly activated and then producing a large number of cytokines and inducing an inflammatory storm. Mesenchymal stem cells (MSCs) have been shown to possess a comprehensive powerful immunomodulatory function. This study aims to investigate the safety and efficacy of intravenous infusion of mesenchymal stem cells in severe patients with COVID-19.

DETAILED DESCRIPTION:
Coronavirus-19 Disease (COVID-19), caused by the Sars-Cov-2 virus, which occurs as a growing pandemic in early 2020 and currently represents an emergency state worldwide. Several reports have shown that the first step in the pathogenesis of Sars-Cov-2 is the recognition of the angiotensin I converting enzyme (ACE2) receptor by the virus. This ACE2 receptor is widely distributed on the surface of human cells, especially as type II alveolar cells and capillary endothelium, however bone marrow, lymph nodes, thymus and spleen are known as immune cells, such as T and lymphocytes. B and macrophages, are negatives to ACE2. These results suggest that immunotherapy can be used to treat infected patients. However, an immunomodulatory capacity cannot be so strong, if just one or two major immunological factors used, as the virus can cause a "cytokine storm", such as IL-2, IL-6, IL-7, GSCF, IP10 , MCP1, MIP1A and TNFα, followed by edema, gas exchange dysfunction, acute respiratory distress syndrome, cardiac injury and secondary infection that can lead to death. Therefore, avoiding a "cytokine storm" may be the key to treating patients infected with Sars-Cov-2. Mesenchymal stem cells (MSCs), due to their potential for immunomodulatory activity, can have beneficial effects in preventing or attenuating the cytokine storm. Because MSCs have been widely used in cell therapy, from basic research to clinical trials. Safety and efficacy have been clearly documented in several clinical trials, especially in immune-mediated inflammatory diseases, such as graft versus host disease (GVHD). The objective of the study is to verify the safety and feasibility of using allogeneic bone marrow mesenchymal stem cells in patients with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmation of COVID19 infection by reverse-transcription polymerase chain reaction (RT-PCR)
* The patient or legal donor agrees to participate in the study and signs the informed consent.
* Patients with orange or red criteria according to the score proposed by Liao et al (2020)

Exclusion Criteria:

* Patient with pregnancy, are planning to become pregnant or breastfeeding
* Patients with malignant blood-borne diseases such as HIV or syphilis
* Not consenting for clinical trial
* Patients with other than orange or red criteria according to the score proposed by Liao et al (2020)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-25 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 60 days
  Assessment of Overall survival at 30 days post intervention

SECONDARY OUTCOMES:
Changes on inflammatory C-reactive protein | 60 days
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of C-reactive protein (mg/dL)
Hospital stay | 60 days
  days of the patients in hospital
Oxygenation index (PaO2/FiO2) | 60 days
  Evaluation of functional respiratory changes: PaO2 / FiO2 ratio
Improvement in Liao's score (2020) | 60 days
  Improvement in Liao's score (2020)
Radiological improvement | 60 days
  Computed tomography Chest assesment will be done to assess improvement in radiological findings of COVID-19
Time of COVID19 PCR negativity | 28 days
  PCR testing to check PCR negativity

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Silla, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: No